CLINICAL TRIAL: NCT00358956
Title: A Phase II, Open-Label Study To Assess The Efficacy and Tolerability of ZD6474 (ZACTIMA™ ) 100 mg Monotherapy In Subjects With Locally Advanced or Metastatic Hereditary Medullary Thyroid Cancer
Brief Title: A Study To Assess ZD6474 (ZACTIMA™) Monotherapy In Locally Advanced or Metastatic Hereditary Medullary Thyroid Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D4200C00068; 2006-001354-28 (EudraCT Number)
Record Dates: First submitted 2006-07-28; First posted 2006-08-01 (Estimated); Results first posted 2012-08-31 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2016-12

CONDITIONS: Thyroid Cancer
Keywords: medullary thyroid cancer; MTC; hereditary medullary thyroid cancer; thyroid cancer
MeSH Terms: conditions — Thyroid Neoplasms; Carcinoma, Medullary; Familial medullary thyroid carcinoma | interventions — vandetanib

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: ZD6474 (vandetanib)

INTERVENTIONS:
Drug: ZD6474 (vandetanib) — 100 mg once daily oral tablet
  Other Names: Caprelsa™

SUMMARY:
This will be a Phase II, open label study to establish the effect of once-daily oral doses of ZD6474 100mg in subjects with locally advanced or metastatic hereditary medullary thyroid cancer in whom no standard therapeutic option is available.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* Previously confirmed histological diagnosis of locally advanced or metastatic hereditary medullary thyroid carcinoma without standard therapeutic options
* Aged 18 or over and a life expectancy of more than 12 weeks

Exclusion Criteria:

* The last dose of prior chemo/radiation received less than 4 weeks before the start of study therapy
* Congenital long QT syndrome or 1st degree relative with unexplained sudden death under 40 years of age, history of arrhythmia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2006-08; Primary Completion 2008-01 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (9):
- United States (2):
  - Research Site, Little Rock, Arkansas
  - Research Site, Boston, Massachusetts
- Research Site, St Leonards, Australia
- Research Site, Sherbrooke, Quebec, Canada
- Research Site, Pisa, Italy
- Research Site, Utrecht, Netherlands
- Research Site, Bucharest, Romania
- Research Site, Madrid, Spain
- Research Site, Basel, Switzerland

REFERENCES:
- [Background] Robinson BG, Paz-Ares L, Krebs A, Vasselli J, Haddad R. Vandetanib (100 mg) in patients with locally advanced or metastatic hereditary medullary thyroid cancer. J Clin Endocrinol Metab. 2010 Jun;95(6):2664-71. doi: 10.1210/jc.2009-2461. Epub 2010 Apr 6. PMID 20371662
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=349&filename=CSR-D4200C00068.pdf
- See also: CSR-D4200C00068.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=349&filename=CSR-D4200C00068.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 29 August 2006 to 31 January 2008, 19 participants in 9 centers in 8 global countries received 100 mg vandetanib.
Pre-assignment Details: 22 participants were screened; 19 participants received treatment.
Groups:
- ZD6474 (ZACTIMA™) 100 mg: ZD6474 (ZACTIMA™)100 mg daily
Period: Overall Study
Arm/Group | ZD6474 (ZACTIMA™) 100 mg
Started | 19
Completed | 11 (ongoing study treatment at data cut-off)
Not Completed | 8
Not completed — Adverse Event | 3
Not completed — condition under investigation worsened | 4
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | ZD6474 (ZACTIMA™) 100 mg
Number analyzed (Participants) | 19
Age, Continuous [Mean (Full Range); unit: years] | 44.7 [22 to 79]
Gender [Count of Participants; unit: Participants]
  Female | 6
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: The ORR is the number of patients that are responders ie those patients with a confirmed best objective response of complete response (CR) or partial response (PR) as defined by RECIST criteria.
  The categories for best objective response are CR, PR, stable disease (SD)>= 12 weeks, progressive disease (PD) or NE.
Time Frame: RECIST assessed at screening (up to 3 weeks prior to first dose), then every 12 weeks (± 2 weeks), from date of first dose to objective progression, up to and including discontinuation of study treatment.
Measure: Number; unit: Participants
Arm/Group | ZD6474 (ZACTIMA™) 100 mg
Number analyzed (Participants) | 19
Participants | 3

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: Median progression free survival (months) estimated from a Weibull model with corresponding 95% confidence intervals. Progression free survival is the time from randomisation until objective disease progression (determined by RECIST assessments) or death (by any cause in the absence of objective progression) provided death is within 3 months from the last evaluable RECIST assessment.
Time Frame: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | ZD6474 (ZACTIMA™) 100 mg
Number analyzed (Participants) | 19
Months | 16.2 [6.8 to 38.6]

3. Secondary Outcome: Disease Control Rate (DCR)
Description: Disease control rate is defined as the number of patients who achieved disease control at 8 weeks following randomisation. Disease control at 8 weeks is defined as a best objective response of complete response (CR), partial response (PR) or stable disease (SD) >= 24 weeks
Time Frame: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | ZD6474 (ZACTIMA™) 100 mg
Number analyzed (Participants) | 19
Participants | 13

4. Secondary Outcome: World Heath Organization (WHO) Performance Status
Description: Number of patients demonstrating an improvement from baseline to 24 weeks in WHO PS. Where WHO PS is the standard scale with patients scored (0 healthy - 5 dead) based on their physical capabilities
Time Frame: WHO PS assessed at screening (up to 3 weeks prior to first dose), baseline and then every 12 weeks (± 2 weeks), up to and including discontinuation of study treatment.
Measure: Number; unit: Participants
Arm/Group | ZD6474 (ZACTIMA™) 100 mg
Number analyzed (Participants) | 19
Participants | 0

5. Secondary Outcome: Symptomatic Response
Description: Symptomatic response will be defined as at least a 50% decrease in the stool frequency (represented by a persistent decrease in stool frequency over 4 weeks), taking as reference the baseline (mean) level.
Time Frame: Symptomatic diarrhea was assessed using stool frequency diaries. Baseline was established using the average of the 4 days immediately prior to first dose, then weekly until discontinuation of study treatment.
Measure: Number; unit: Participants
Arm/Group | ZD6474 (ZACTIMA™) 100 mg
Number analyzed (Participants) | 19
Participants | 0

6. Secondary Outcome: Biochemical Response Calcitonin (CTN )
Description: A patient's best biochemical response was calculated from assessments performed at baseline and during treatment. Responders were those patients with a best biochemical response of CR or PR, confirmed by repeat assessments, which were to be performed no less than 4 weeks after the criteria for PR or CR were first met.
Time Frame: Blood samples for analysis of CTN were taken at screening (0, 1, 4, and 8 hours to determine the baseline CTN/CEA level) then every 4 weeks until discontinuation Time point(s) at which outcome measure was assessed. (Limit: 255 characters)
Measure: Number; unit: Participants
Arm/Group | ZD6474 (ZACTIMA™) 100 mg
Number analyzed (Participants) | 19
Participants | 3

7. Secondary Outcome: Biochemical Response Carcinoembryonic Antigen CEA)
Description: A patient's best biochemical response was calculated from assessments performed at baseline and during treatment. Responders were those patients with a best biochemical response of CR or PR, confirmed by repeat assessments, which were to be performed no less than 4 weeks after the criteria for Partial Response (PR) or Complete Response (CR) were first met.
Time Frame: Blood samples for analysis of CTN were taken at screening (0, 1, 4, and 8 hours to determine the baseline CTN/CEA level) then every 4 weeks until discontinuation
Measure: Number; unit: Participants
Arm/Group | ZD6474 (ZACTIMA™) 100 mg
Number analyzed (Participants) | 19
Participants | 1

ADVERSE EVENTS:
Arm/Group | ZD6474 (ZACTIMA™) 100 mg
Serious Adverse Events (participants affected / at risk) | 4/19
Other Adverse Events (participants affected / at risk) | 18/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ZD6474 (ZACTIMA™) 100 mg (N=19)
Diabetes Insipidus (Endocrine disorders) | 1
Phaeochromocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ZD6474 (ZACTIMA™) 100 mg (N=19)
Deafness Unilateral (Ear and labyrinth disorders) | 1
Hypothyroidism (Endocrine disorders) | 2
Conjunctivitis (Eye disorders) | 1
Diplopia (Eye disorders) | 1
Visual Disturbance (Eye disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 9
Constipation (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 3
Abdominal Pain (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 2
Flatulence (Gastrointestinal disorders) | 2
Dry Mouth (Gastrointestinal disorders) | 1
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Oral Discomfort (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 9
Asthenia (General disorders) | 2
Influenza Like Illness (General disorders) | 1
Malaise (General disorders) | 1
Mucous Membrane Disorder (General disorders) | 1
Thirst (General disorders) | 1
Folliculitis (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 1
Furuncle (Infections and infestations) | 1
Paronychia (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Tinea Pedis (Infections and infestations) | 1
Upper Respiratory Tract Infection (Infections and infestations) | 1
Weight Decreased (Infections and infestations) | 2
Electrocardiogram Qt Prolonged (Infections and infestations) | 1
Weight Increased (Infections and infestations) | 1
Anorexia (Metabolism and nutrition disorders) | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Mobility Decreased (Musculoskeletal and connective tissue disorders) | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 1
Dysarthria (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 2
Mood Altered (Psychiatric disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Renal Failure (Renal and urinary disorders) | 1
Erectile Dysfunction (Reproductive system and breast disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1
Upper Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 5
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 3
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 2
Dry Skin (Skin and subcutaneous tissue disorders) | 2
Acne (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Purpura (Skin and subcutaneous tissue disorders) | 1
Rash Erythematous (Skin and subcutaneous tissue disorders) | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 3
Flushing (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.